CLINICAL TRIAL: NCT04259710
Title: Pedometer Program:Every Step Counts
Brief Title: Do Implementation Intentions Increase Average Daily Step Count.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Donna R Zwas, Senior Cardiologist, Hadassah Medical Organization
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: HMO0523-18
Record Dates: First submitted 2019-12-04; First posted 2020-02-06 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Stage 1: Comparison of intervention groups to pedometer only group. Stage 2: Comparison of intervention with implementation intentions to intervention alone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pedometer only (Placebo Comparator): participants will be given a pedometer and instructed how to use it, but will not participate in the goal setting intervention.
  Interventions: Behavioral: Pedometer only
- Pedometer and intervention (Active Comparator): participants will be given a pedometer and participate in a weekly goal setting meeting with the investigator and will receive weekly tips.
  Interventions: Behavioral: Goal-setting intervention
- Pedometer, intervention and implementation intentions (Experimental): participants will be given a pedometer and participate in the weekly goal setting as above. In addition, 3 times during the intervention they will fill out a form that encourages performance of implementation intentions.
  Interventions: Behavioral: Goal-setting intervention; Behavioral: Goal setting with implementation intentions

INTERVENTIONS:
Behavioral: Goal-setting intervention — The participant will meet weekly with the investigator, report steps and set goals for the following week.
  Arms: Pedometer and intervention; Pedometer, intervention and implementation intentions
Behavioral: Goal setting with implementation intentions — In addition to the standard goal-setting intervention, the participant will fill out a form that directs them to perform implementation intentions at weeks 1, 5 and 9.
  Arms: Pedometer, intervention and implementation intentions
Behavioral: Pedometer only — the participant will be given a pedometer and instructed how to use it.
  Arms: Pedometer only

SUMMARY:
Cardiovascular disease is the second major cause of death for women in Israel and the leading cause of death among women worldwide. Women have higher mortality rates after a coronary or cerebrovascular event compared to men, and receive less attention for prevention and treatment of heart disease.

The risk factors for heart disease among women in Israel are high: 53% of women in the State of Israel are overweight or obese and 48% of women do not exercise.

Increasing physical activity can lower the risk of developing cardiovascular disease in women. The literature suggests that even minor changes in behavior can reduce the morbidity, mortality and costs to the health care system.

Pedometers have proven to be an effective tool for increasing physical activity, and have the potential to create change in health habits. The pedometer measures steps and is a simple measure that gives an estimate of the extent of exercise in terms of steps. The device is simple and user-friendly and serves as an indicator of movement as a result of health choices. The literature shows that when pedometers are integrated into a support program, they provide an incentive to increase physical activity. Supporting software includes, among other things - choosing personal goals, close tracking, and self-tracking and re balancing systems. "Implementation intention" is a strategy in the form of an "if-then plan" that can increase the likelihood of attaining one's goals. It is different than specifying a goal intentions as it specifies the when, where and how portions of goal-directed behavior. This study seeks to compare the increase in steps in participants randomly assigned in a 2:2:1 allocation to a goal-setting pedometer intervention, a goal-setting plus implementation intentions pedometer intervention vs pedometer only.

DETAILED DESCRIPTION:
Goals-

1. Increasing step count as measured by a pedometer in hospital employees. The overall goal is for each participant to reach 10,000 steps a day at the end of the 12 weeks of intervention.
2. Comparison of increase in steps in participants who undergo an implementation intentions intervention in addition to a goal setting intervention to those who receive the goal setting intervention alone, to those assigned to pedometer without goal setting intervention. The goal setting intevention includes setting weekly goals with the investigator, and receiving weekly tips.

   The implementation intention group will fill out an action planning form 3 times during the course of the intervention.

   The pedometer only group will receive a pedometer and instructions as to it's use.
3. Examining the effect of self-efficacy on increasing the amount of steps among program participants.
4. Examining the effect of the program on a measure of burnout in the workplace among program participants.
5. Examining the impact of a program designed to increase physical activity (through walking) on self-report of nutrition behavior.
6. Examining the correlation between emotional self-regulation as measured on a self-report measure and success in increasing steps.
7. Examining the effect of the program on physiological measures: BMI, blood pressure, pulse, and waist circumference.

Target population- Hadassah Medical Center employee and volunteers

sample size- 180 Hadassah employee and volunteers to be enrolled in the program, using the first to enroll method. The sample size was calculated based on an expected 1000 step difference between the intervention groups with implementation intentions vs the group without implementation intentions. change in the number of steps per day between the control group and the intervention groups, as shown in previous studies. Under a 2350 Sd assumption, a sample size of 87 participants in each group would provide a power of 80% to detect a 5% significance level change.

ELIGIBILITY:
Inclusion Criteria:

* Hadassah employees, volunteers and retirees
* able to commit to 12 week program
* no medical contraindication to physical activity

Exclusion Criteria:

* unable to walk
* unable to maintain and use the pedometer
* unable to provide informed consent

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — participant eligibility is based on self-representation of gender identity.
Enrollment: 280 (Estimated)
Dates: Start 2014-10-21 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Step count | 13 weeks
  Average step count over 5 days of the last week of participation in the protocol

SECONDARY OUTCOMES:
Blood pressure | 13 weeks
  systolic and diastolic blood pressure at final visit
Body mass index | 13 weeks
  weight and height will be combined to report BMI in kg/m^2
waist circumference | 13 weeks
  cm
Percentage increase in steps | 13 weeks
  (average daily steps on final visit) - (average daily steps on first visit)/(average daily steps on first visit)
self report of burnout | 13 weeks
  Shiron-Melamed burnout questionnaire 14 item scale, scores range from 14 to 98 with higher scores reflecting more burnout
resting heart rate | 13 weeks
  heart rate measured over 60 seconds at rest
physical activity self efficacy | 13 weeks
  Schwarzer physical activity self efficacy scale, range 4-20, higher score = higher self efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Donna R Zwas, MD MPH, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel